CLINICAL TRIAL: NCT02780323
Title: A Multi-center, Double-blind, Active-controlled, Randomized, Parallel-group Clinical Trial to Compare the Efficacy and Safety of CELBESTA® and CELEBREX® in Patients With Rheumatoid Arthritis
Brief Title: Study to Compare the Efficacy and Safety of CELBESTA® and CELEBREX® in Patients With Rheumatoid Arthritis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dong-A ST Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CELB_RA_IV
Record Dates: First submitted 2016-05-19; First posted 2016-05-23 (Estimated); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Rheumatoid Arthritis
Keywords: Celecoxib; CELBESTA
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Celecoxib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- CELBESTA® and CELEBREX® placebo (Experimental): CELBESTA® and CELEBREX® placebo is administered twice daily for 6 weeks
  Interventions: Drug: CELBESTA®; Drug: CELEBREX® placebo
- CELEBREX® (Active Comparator): CELEBREX® and CELBESTA® placebo is administered twice daily for 6 weeks
  Interventions: Drug: CELEBREX®; Drug: CELBESTA® placebo

INTERVENTIONS:
Drug: CELBESTA® — 1 tablet of CELBESTA® and 1 tablet of CELEBREX® placebo, twice daily for 6 weeks
  Other Names: celecoxib
  Arms: CELBESTA® and CELEBREX® placebo
Drug: CELEBREX® — 1 tablet of CELEBREX® and 1 tablet of CELBESTA® placebo, twice daily for 6 weeks
  Other Names: celecoxib
  Arms: CELEBREX®
Drug: CELEBREX® placebo — 1 tablet of CELBESTA® and 1 tablet of CELEBREX® placebo, twice daily for 6 weeks
  Other Names: celecoxib placebo
  Arms: CELBESTA® and CELEBREX® placebo
Drug: CELBESTA® placebo — 1 tablet of CELEBREX® and 1 tablet of CELBESTA® placebo, twice daily for 6 weeks
  Other Names: celecoxib placebo
  Arms: CELEBREX®

SUMMARY:
This Phase IV clinical study is to Compare the Efficacy and Safety of CELBESTA® and CELEBREX® in Rheumatoid Arthritis Patients

DETAILED DESCRIPTION:
Thisi is a multi-center, double-blind, active-controlled, randomized, parallel-group clinical trial to compare the efficacy and safety of CELBESTA® and CELEBREX® in patients with rheumatoid arthritis. The subject will receive two tablets twice daily for 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Anyone over the age of 19
* Subjects who are diagnosed as established rheumatoid arthritis at screening visit and before
* Pain greater than 40/100mm-VAS(Visual Analgue Scale) after wash-out period
* Patients who are taking oral corticosteroids without dosage change (within a range of prednisolone 10mg a day) at least 4weeks and more than 1 DMARDs at least 3 months from screening test
* Patients willing and able to provide signed informed consent after the nature of the study has been explained

Exclusion Criteria:

* History of angina pectoris or congestive heart failure at rest or minimum activity
* History of myocardial infarction or artherosclerosis
* Patients who had a coronary angioplaty or coronary artery bypass graft within 1 year
* History of stroke, transient ischemic attack or hepatitis within 2 years
* Patients who have uncontrolled hypertension at screening
* Patients who take the medicines that might effect the test results by study investigators or might cause a excessive risk to the patients

  * Intra-articular corticosteroid injection within 4 weeks from screening
  * biological DMARDs such as infliximab, adlimumab, entanercept, anakinara or abatacept wihin 6 months from randomization
  * biological DMARDs such as rituximab within 1 year from randomization
* History of a malignant tumor (except for the patients whose tumor was removed and there's no recurrence within 5 years)
* Patients who have gastrointestinal bleeding or peptic ulcer (except scar) within 30 days
* History of a gastroesophageal surgery such as antigastric-secretion surgery or esophagogastrectomy (except a simple perforator surgery)
* Patients who have severe disability in GI, Kidney, Liver and Blood
* Pregnant women, Lactating women and Women of child-bering potential who are not using adequate means of contraception
* History of allergy to COX-2 inhibitors or sulphonamides or other NSAIDs
* Any condition that, in the view of the investigator, would interfere with study participation

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2015-11-02 (Actual); Primary Completion 2017-12-26 (Actual); Study Completion 2017-12-26 (Actual)

PRIMARY OUTCOMES:
Change from baseline of 100mm VAS about pain in study at week 6 | week 6

SECONDARY OUTCOMES:
Change from baseline of DAS28-ESR(Disease Activity Score in 28 joints) at week 6 | week 6

CONTACTS AND LOCATIONS:
Overall Officials: Seung-jae Hong, MD,PhD, Principal Investigator — Kyung Hee University Hospital; Sungsoo Kim, MD,PhD, Principal Investigator — Gangneung Asan Hospital; Sangil Lee, MD,PhD, Principal Investigator — Gyeongsang National Hospital; Changnam Son, MD,PhD, Principal Investigator — Keimyung University Dongsan Medical Center; Yeong Ho Seo, MD,PhD, Principal Investigator — Korea University; Geun-Tae Kim, MD,PhD, Principal Investigator — Kosin University Gospel Hospital; Jin-Wuk Hur, MD,PhD, Principal Investigator — Seoul Eulji Hospital; Hyun-Sook Kim, MD,PhD, Principal Investigator — Soonchunhyang University Hospital; Myeong Soo Lee, MD,PhD, Principal Investigator — Wonkwang University Hospital; Yun Sung Kim, MD,PhD, Principal Investigator — Chosun University Hospital
Locations (1):
- Kyung Hee University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No